CLINICAL TRIAL: NCT03571230
Title: 10-Day Antimicrobial Susceptibility Testing Guided Triple Therapy Versus 14-Day Empirical Tailored Therapy for the First-line Treatment of Helicobacter Pylori Infection-A Randomized Controlled Trail
Brief Title: Antimicrobial Susceptibility Testing Guided Therapy Versus Empirical Therapy for the First-line Helicobacter Pylori Eradication.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017SDU-QILU-G003
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori Infection; Antimicrobial Susceptibility Testing
Keywords: Helicobacter Pylori Infection; Antimicrobial Susceptibility testing(AST)
MeSH Terms: interventions — Clarithromycin; Metronidazole; Tinidazole; Levofloxacin; Furazolidone; Tetracycline

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Antimicrobial susceptibility testing guided therapy (Experimental): Patients in this group will receive a 10-day triple therapy for the Helicobacter pylori eradication. The regimen contains one proton pump inhibitor and two sensitive antibiotics determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline will be evaluated.
  Drugs: 1.one proton pump inhibitor: lansoprazole 30mg bid for 10d 2.two sensitive antibiotics: amoxicillin 1000mg bid for 10d, clarithromycin 500mg bid for 10d, metronidazole 500mg tid for 10d, tinidazole 500mg tid for 10d, levofloxacin 500mg qd for 10d, furazolidone 100mg bid for 10d, tetracycline 750mg bid for 10d.
  Interventions: Drug: two sensitive antibiotics(amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline); Drug: one proton pump inhibitor(PPI)
- Empirical tailored therapy (Experimental): Patients in this group will receive a 14-day bismuth-based quadruple therapy for the H.pylori eradication. The regimen contains one PPI, Colloidal Bismuth Pectin and two antibiotics based on personal medication history. If the patient has taken clarithromycin, roxithromycin and azithromycin for less than 2 weeks before, he will be treated with amoxicillin and clarithromycin. Otherwise, he will be treated with amoxicillin and furazolidone.
  Drugs: 1.one proton pump inhibitor: lansoprazole 30mg bid for 14d 2.Colloidal Bismuth Pectin 200mg bid for 14d 3.two antibiotics based on personal medication history: amoxicillin 1000mg bid and clarithromycin 500mg bid for 14d, amoxicillin 1000mg bid and furazolidone 100mg bid for 14d.
  Interventions: Drug: two antibiotics based on personal medication history(amoxicillin,clarithromycin,furazolidone); Drug: one proton pump inhibitor(PPI); Drug: Colloidal Bismuth Pectin
- Salvage therapy for negative culture (Other): When the culture results are negative, patients will receive 14-day empirical tailored therapy based on personal medication history.
  Drugs: 1.one proton pump inhibitor: lansoprazole 30mg bid for 14d 2.Colloidal Bismuth Pectin 200mg bid for 14d 3.two antibiotics based on personal medication history: amoxicillin 1000mg bid and clarithromycin 500mg bid for 14d, amoxicillin 1000mg bid and furazolidone 100mg bid for 14d.
  Interventions: Drug: two antibiotics based on personal medication history(amoxicillin,clarithromycin,furazolidone); Drug: one proton pump inhibitor(PPI); Drug: Colloidal Bismuth Pectin
- Salvage therapy for failed eradication (Other): If patients failed with AST guided eradication therapy or empirical therapy, patients will be treated with another 14-day bismuth-based quadruple therapy.
  Drugs: 1.one proton pump inhibitor: lansoprazole 30mg bid for 14d 2.Colloidal Bismuth Pectin 200mg bid for 14d 3.two antibiotics for rescue therapy: tetracycline 750mg bid and furazolidone 100mg bid for 14d.
  Interventions: Drug: one proton pump inhibitor(PPI); Drug: Colloidal Bismuth Pectin; Drug: two antibiotics for failed eradication(tetracyclin,furazolidone)

INTERVENTIONS:
Drug: two sensitive antibiotics(amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline) — Patients will receive a 10-day triple therapy for the H.pylori eradication. The regimen contains one PPI and two sensitive antibiotics determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline will be evaluated.
  Arms: Antimicrobial susceptibility testing guided therapy
Drug: two antibiotics based on personal medication history(amoxicillin,clarithromycin,furazolidone) — Patients will receive a 14-day bismuth-based quadruple therapy for the H.pylori eradication. The regimen contains one PPI, Colloidal Bismuth Pectin and two antibiotics based on personal medication history. If the patient has taken clarithromycin, roxithromycin and azithromycin for less than 2 weeks before, he will be treated with amoxicillin and clarithromycin. Otherwise, he will be treated with amoxicillin and furazolidone.
  Arms: Empirical tailored therapy; Salvage therapy for negative culture
Drug: one proton pump inhibitor(PPI) — All the patients need this drug.
Drug: Colloidal Bismuth Pectin — All the patients treated with 14-day bismuth-based quadruple therapy need this drug.
  Arms: Empirical tailored therapy; Salvage therapy for failed eradication; Salvage therapy for negative culture
Drug: two antibiotics for failed eradication(tetracyclin,furazolidone) — If the patients failed with AST guided eradication therapy or empirical therapy, patients will be treated with another 14-day bismuth-based quadruple therapy. The regimen contains one PPI, Colloidal Bismuth Pectin, tetracycline and furazolidone.
  Arms: Salvage therapy for failed eradication

SUMMARY:
The purpose of this study is to assess efficacy of 10-day antimicrobial susceptibility test guided triple therapy for the first-line treatment of Helicobacter pylori infection, then comparing it with 14-day empirical tailored therapy to tell which one has a better performance in both efficacy and safety.

DETAILED DESCRIPTION:
Helicobacter pylori(H.pylori), which infects about 50% of the global population, has been recognized as a main risk factor of multiple gastric pathologies, especially non-cardiac gastric cancer. Strongly evidence supports that H.pylori eradication is an effective approach to reduce the incidence of those pathologies. Antimicrobial susceptibility test can pick out sensitive drugs to kill Helicobacter pylori, and reduce secondary drug resistance. But, there is a lack of high quality RCT to compare its efficacy with empirical regimen in the first-line treatment.

Our study aims to assess the efficacy of 10-day antimicrobial susceptibility test guided triple therapy for the first-line treatment of Helicobacter pylori infection. Comparing this regimen with 14-day Empirical Tailored Therapy to tell which one is better in clinic practice. We also want to find whether the 10-day antimicrobial susceptibility test guided triple therapy has less intestinal dysbacteriosis with a shorter duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with H. pylori infection.

Exclusion Criteria:

* Patients with previous H. pylori eradication therapy;
* Patients unable or unwilling to receive gastroscopy;
* Patients treated with H2-receptor antagonist, PPI, bismuth and antibiotics in the previous 4 weeks;
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Patients with known or suspected allergy to study medications;
* Currently pregnant or lactating;
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rates in 2 groups | 6 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rate of improving dyspepsia symptoms after Helicobacter pylori eradication. | 6 months
  Dyspepsia symptoms will be measured using a 8-point Likert scale, and patients rate their symptoms from 0 (none) to 8 (severe) before and after the Helicobacter pylori eradication.
The rate of adverse events happening | 6 months
  Similarly, adverse events will also be measured by the Likert scale.
The rate of good compliance | 6 months
  Patients taken over 90% of drugs are considered to have a good compliance.
Difference of cost per patient for each eradication achieved in two groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Xiuli Zuo, Jinan, Shandong, China